CLINICAL TRIAL: NCT06240039
Title: Direct Versus Indirect Effect of Amino Acids on Hepatokines in Healthy Subjects and Patients With Non-alcoholic Fatty Liver Disease
Brief Title: Direct Versus Indirect Effect of Amino Acids on Hepatokines
Acronym: Diaakine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Nicolai Jacob Wewer Albrechtsen, Associate Professor, MD, PhD, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Diaakine
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluating the direct and indirect effect of amino acids on the regulation of hepatokines (Experimental): Participants will be subjected to four experimental days
  Interventions: Other: Evaluating the acute effect of an amino acid infusion with and without a concomitant infusion of the somatostatin analogue octreotide to eliminate endogenous production of glucagon

INTERVENTIONS:
Other: Evaluating the acute effect of an amino acid infusion with and without a concomitant infusion of the somatostatin analogue octreotide to eliminate endogenous production of glucagon — The experimental days consist of four study days:
  1. Assessment of liver fat and visceral fat by magnetic resonance imaging (MRI; 6-point Dixon) (study day A)
  2. Somatostatin infusion (4 hours) plus amino acid infusion (45 minutes) (study day B)
  3. Saline infusion (4 hours) plus amino acid infusion (45 minutes) (study day C)
  4. Somatostatin infusion (4 hours) plus saline infusion (45 minutes) (study day D)
  The subjects will participate in the experimental days (study day B to D) in randomized order on three different days. For study day B to D, at timepoint t = -75, subjects will receive either; a 240-minute intravenous infusion of a somatostatin analogue (at 200 ng/kg/min (infusion rate will not exceed 1000 µg/hour) or saline. After 75 minutes (timepoint t = 0), the subjects will receive a 45-minute intravenous infusion of amino acids or saline at 3.885 ml/kg/hour.
  In total, blood will be sampled 11 times over a period of 6 hours and 15 minutes.

SUMMARY:
Liver hormones are key metabolic regulators and increased in metabolic diseases, including fatty liver disease. The underlying mechanisms driving the elevated levels are currently unknown and presents a major challenge in understanding the interplay between liver hormones and fatty liver disease. The project aims to investigate what stimulates the liver to secrete its hormones and why the secretion is increased in patients with fatty liver disease. The investigator (Associate Prof. Nicolai J Wewer Albrechtsen) will investigate the direct and indirect effects of an amino acid amino infusion on the secretion of hepatokines in individuals with and without metabolic dysfunction-associated steatotic liver disease (MASLD).

DETAILED DESCRIPTION:
The liver secretes signaling molecules, (termed hepatokines) to the blood circulation which are powerful metabolic regulators and biomarkers of liver disease. Some of the more studied hepatokines include follistatin, fibroblast growth factor 21 (FGF21) and growth differentiation factor 15 (GDF15) and they have been sown to improve glucose tolerance, reduce liver fat content and regulate appetite.

In dysregulated metabolic conditions, including obesity, MASLD and type 2 diabetes, the circulating levels of hepatokines are increased. It could be speculated that the body increases hepatokine levels as a feedback mechanism to combat dysregulated metabolism. However, the underlying mechanisms driving the elevated levels in metabolic disease are currently unknown. The secretion of follistatin, FGF21 and GDF15 from the liver has been suggested to be stimulated by glucagon and amino acids. In dysregulated metabolic diseases, circulating levels of glucagon and amino acids are often increased and are highly dependent on hepatic steatosis. Increased levels of hepatokines observed in dysregulated metabolic individuals could therefore be attributed to an increase in circulating glucagon, amino acids, or a combination of both.

The study aims to explore the direct and indirect effect of amino acids on the regulation of hepatokines in individuals with and without MASLD. The study evaluates the acute effect of an amino acid infusion with and without a concomitant infusion of the somatostatin analogue octreotide to eliminate endogenous production of glucagon, thus isolating the direct effect of amino acids. ,

The investigators hypothesizes that an amino acid infusion will increase the secretion of hepatokines independent of glucagon.

ELIGIBILITY:
Group 1: (Lean controls)

Inclusion Criteria:

* Male or female between 25-65 years of age at time of screening
* Body mass index of 18.6-25 kg/m2

Exclusion Criteria:

* Contraindications for MRI-scan
* Severe liver disease (estimated by FIB4 score > 3.25)
* Type 2 diabetes according to ADA criteria
* Significant history of alcoholism or drug/chemical abuse as per investigators judgement
* Amino acid related diseases
* Kidney disease
* Cardiac problems
* Cancer within the past 1 year
* Anemia
* Pregnancy or breast feeding
* Smoking
* Any medicine, acute illness (within the last two weeks) or other circumstances that in the opinion of the investigator might endanger the participants' safety or compliance with the protocol

Group 2 (individuals with hepatic steatosis):

Inclusion Criteria:

* Male or female between 25-65 years of age at time of screening
* Body mass index of 25-40 kg/m2
* Hepatic non-alcoholic steatosis verified by liver biopsy, fibroscan or ultrasound

Exclusion Criteria:

* Contraindications for MRI-scan
* Severe liver disease (estimated by FIB4 score > 3.25)
* Type 2 diabetes according to ADA criteria
* Significant history of alcoholism or drug/chemical abuse as per investigators judgement
* Amino acid related diseases
* Kidney disease
* Cardiac problems
* Cancer within the past 1 year
* Anemia
* Pregnancy or breast feeding
* Smoking
* Any medicine, acute illness (within the last two weeks) or other circumstances that in the opinion of the investigator might endanger the participants' safety or compliance with the protocol

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The direct (amino acid + somatostatin) versus the indirect (amino acid + placebo) effect of amino acids on circulating levels of follistatin. | From blood sample at minute 0 until blood sample at minute 300.
  Defined as the difference in incremental AUC0-300 min (iAUC) of follistatin between study day B and study day C in healthy individuals.

SECONDARY OUTCOMES:
The direct (amino acid + somatostatin) versus the indirect (amino acid + placebo) effect of amino acids on circulating levels of FGF21 and GDF15 | From blood sample at minute 0 until blood sample at minute 300.
  Defined as the difference in iAUC0-300 min between study day B and study day C in healthy individuals.
The direct versus the indirect effect of amino acids on circulating levels of hepatokines (follistatin, FGF21 and GDF15). | From blood sample at minute 0 until blood sample at minute 300
  Defined as the difference in iAUC0-300 min of hepatokines between study day B and study day C in individuals with MASLD.
Differences between healthy and MASLD in the increase in hepatokines during study day B (direct effect of amino acids) | From blood sample at minute 0 until blood sample at minute 300
  Defined as the differences in iAUC0-300 min of hepatokines between healthy and MASLD
Differences between healthy and MASLD in the increase in hepatokines during study day C (indirect effect of amino acids). | From blood sample at minute 0 until blood sample at minute 300
  Defined as the differences in iAUC0-300 min of hepatokines between healthy and MASLD
The inhibitory effect of somatostatin versus the stimulatory effect of amino acids on glucagon, insulin and C-peptide levels during study day B in healthy and MASLD. | From blood sample at minute -75 until blood sample at minute 45
  Defined as the difference between iAUC -75-0 min and iAUC0-45 min in both groups
Differences in glucagon, insulin and C-peptide concentrations between study day B and C in healthy and MASLD | From blood sample at minute 0 until blood sample at minute 300
  Defined as the difference between iAUC0-300 min during study day B and C in healthy and MASLD

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
We have not decided to share IPD as this also would require approval from the ethical and data approval committee.